CLINICAL TRIAL: NCT05717205
Title: Pathophysiology of Diabetic Gastroparesis
Acronym: PATODIAG
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Hvidovre University Hospital (Other)
Collaborators: Zealand University Hospital (Other); Steno Diabetes Center Copenhagen (Other)
Responsible Party: Principal Investigator, Melina Svraka Hansen, Principal Investigator, Hvidovre University Hospital
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: SJ-980
Record Dates: First submitted 2022-12-12; First posted 2023-02-08 (Actual); Last update posted 2023-04-14 (Actual); Status verified 2023-04

CONDITIONS: Gastroparesis Due to Diabetes Mellitus Type I
Keywords: gastroparesis
MeSH Terms: conditions — Gastroparesis | interventions — Gastroscopy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- cases with gastroparesis (Active Comparator): patients with a gastroparesis symptom score index (GCSI) of > 1.9 will be considered as cases with gastroparesis and will be subjected to technetium-scintigraphy and gastroscopy with tissuesamples from antrum and fundus and bloodsamples of glucosemetabolism
  Interventions: Diagnostic Test: technetium scitigraphy
- Controls without gastroparesis (Active Comparator): patients with a gastroparesis symptom score index (GCSI) of < 1.9 will be considered as controls without gastroparesis and will be subjected to technetium-scintigraphy and gastroscopy with tissuesamples from antrum and fundus and bloodsamples of glucosemetabolism
  Interventions: Diagnostic Test: technetium scitigraphy

INTERVENTIONS:
Diagnostic Test: technetium scitigraphy — patients will have a technetium scintraphy confirming or ruling out gastroparesis. Then the patients will have a gastroscopy with tissue samples from antrum and fundus. During gastroscopy an endo-flip ballon will meassure the distensibility in pylorus.
  Other Names: gastroscopy with tissuesamples

SUMMARY:
The goal of this study is to explore the pathophysiology of diabetic gastroparesis by conducting an exploratory cohort study. Participants will be type 1 diabetes patients with and without gastroparesis. Investigators will investigate

* Differences in nervefiber density and morphology
* Cellular and transcriptional changes and indices of glucosemetabolism between groups

DETAILED DESCRIPTION:
Aims To perform an exploratory cohort study including 26 type 1 diabetes (DM1) patients aged 18-85 years with gastroparesis and 26 comparable DM1 diabetes patients without gastroparesis, investigating nerve fibre density and length in the mucosal and submucosal layer of the stomach (fundus, and antrum). A variety of molecular, biochemical and cellular experimental procedures will be performed on bloodsamples and tissue biopsies collected during gastroscopy exploring the pathophysiology of gastroparesis. In addition, we will compare differences in, measures of glucose metabolism in the two patient groups through bloodsamples.

Hypotheses

1. Nerve fibre morphology in the stomach is different in type 1 diabetes patients with diabetic gastroparesis compared to diabetes patient without gastroparesis and associated with differences in glucose metabolism and the severity of autonomic and peripheral neuropathy.
2. Patients with gastroparesis show loss of interstitial cells of Cajal (ICC) in the gastric body, antrum and fundus and have marked morphological changes indicative of injuries.
3. Macrophages are thought to play a central role in diabetic gastroparesis, in which a loss of anti-inflammatory heme-oxygenase-1 (HO-1) positive macrophages leads to decreased protection against oxidative stress, resulting in damage to ICCs.
4. In gastroparesis there is increased presence of fibrosis in the stroma and alteration in inflammatory cells.
5. Patients with gastroparesis may have decreased levels of neurotransmitters such as NO and substance P.
6. Gastroparesis may cause pathological alterations of enteric glial and ganglion cells and the cytoplasm of smooth muscle cells.
7. Patients with gastroparesis have lower pyloric distensibility.
8. Examining transcriptional changes in between groups will reveal new genes associated with disease development. Newly developed in vitro models make it possible to explore and correlate molecular biochemical and cellular factors to disease development and progression.

Study Design All participants will be type 1 diabetes patients attending treatment at Steno Diabetes Center Copenhagen (SDCC) or type 1 diabetes patients referred from other treatment facilities. Patients will fill out the Gastroparesis Cardinal Symptom Index (GCSI) questionnaire and be asked if they have been diagnosed with gastroparesis. Patients with known gastroparesis or with a GCSI score ≥ 1.9 without known gastroparesis will be subject to a technetium scintigraphy. Patients without established gastroparesis and a GCSI score < 1.9 will also undergo technetium scintigraphy. A gastric content above 10%, 4 hours after meal ingestion will be considered the diagnostic threshold for gastroparesis Patients with gastroparesis will be considered as cases and patients without gastroparesis as control. All patients will have a gastroscopy to rule out other causes to gastro-intestinal symptoms. During gastroscopy, 8 biopsies will be obtained and endo-flip will be used to measure distesibility in pylorus. Tissue specimens and blood samples will be collected and used in various research-based analyses to understand the pathophysiology.

ELIGIBILITY:
Inclusion Criteria:

* Type 1 diabetes
* age 18-85
* Case group: Gastroparesis verified by technetium scintigraphy and a GCSI score ≥ 1.9
* Control group: Gastroparesis not confirmed by technetium scintigraphy and score GCSI score < 1.9

Exclusion Criteria:

* Ongoing cancer treatment or other concurrent illness that will make the patient unable to attend the study on the discretion of the investigator.
* Recent gastrointestinal surgery
* Active duodenal/gastric ulcer disease,
* Diseases in the ventricle or previously complicated upper abdominal surgery
* Pregnancy or breast feeding
* Persons who, in the judgement of the investigator, may be unable to follow the protocol.
* Parkinson disease
* metoclopramide 48 hours prior to scintigraphy
* domperidone 48 hours prior to scintigraphy
* macrolide antibiotics 48 hours prior to scintigraphy
* anti-cholinergic agents
* Tricycliv antidepressants
* Glucagon-like peptide-1 analogues
* Lithium
* Diphenhydramine
* dopamine agonists
* progesterone, L-dopa
* calcitonine
* ocreotide
* Interferon alfa
* sucralsulfate
* botulinum toxin injections (eg, Botox®) by pyloric injection.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 52 (Estimated)
Dates: Start 2023-02-16 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2025-06-01 (Estimated)

PRIMARY OUTCOMES:
mucosal nerve length density (MNLD) | 24 months
  differences in mucosal nerve length density (MNLD) of the gastric fundus and antrum in diabetes patients with and without gastroparesis. MNLD will be assessed by confocal microscopy of mucosal biopsies obtained by oesophago-gastro-duodenoscopy.

SECONDARY OUTCOMES:
Nerve fibre morphology | 24 months
  Nerve fibre morphology assessed by confocal microscopy of mucosal biopsies obtained by esophago-gastro-duodenoscopy
Differences in histology | 24 months
  Hematoxylin and eosin (HE) staining and c-KIT staining of immune cells, interstitial cells, glia cells, ganglion cells and smooth muscle cells and visualization under a microscope
Transcriptional changes | 24 months
  Altered transcriptional changes in mRNA by NanoString.
Differences in cell populations | 24 months
  Differences in cell populations by fluorescence-activated cell sorting (FACS).
Differences in pyloric distensibility | 24 months
  Pyloric distensibility measurements by Endo-Flip.
Differences in glucose metabolism | 24 months
  plasma glucose in mmol/L, HbA1c in mmol/mol, proinsulin C-peptide in pmol/L
Differences in gastric emptying time | 24 months
  Gastric emptying time assessed by technetium scintigraphy.
Differences in neuropathy measures | 24 months
  sensory tests that record sensation of touch, vibration, cooling and heat.
Immunohistochemical differences | 24 months
  Immunohistochemical staining that uses antibodies to visualize the localization of particular proteins within single cells.

CONTACTS AND LOCATIONS:
Overall Officials: Melina S Hansen, MD, Principal Investigator — Copenhagen University Hospital, Hvidovre
Locations (1):
- Hvidovre University Hospital, Hvidovre, Capital Region, Denmark

IPD SHARING:
Plan to Share IPD: No